CLINICAL TRIAL: NCT07129265
Title: Countering E-cigarette Marketing in the Retail Environment Among Adolescents and Young Adults
Brief Title: Understanding Vape Marketing Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Dana-Farber/Harvard Cancer Center (DF/HCC) Boston, MA (Unknown)
Responsible Party: Principal Investigator, Shivani Gaiha, Faculty Researcher, Boston Children's Hospital
Other Study IDs: 25-232; 5R00CA267477 (NIH)
Record Dates: First submitted 2025-08-05; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: E-cigarette; Vaping; Tobacco; Nicotine; Adolescent Behavior; Video Information; Digital Education Interventions
Keywords: e-cigarette; vaping; tobacco; nicotine; adolescent; counter-marketing; digital content; digital education interventions
MeSH Terms: conditions — Vaping; Adolescent Behavior | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Working group members: 10 members of the expert working group: 2 middle school students, 2 high school students, 2 young adults, 1 educator, 1 parent, and 4 curriculum design expert
  Interventions: Other: Working group
- Focus group participants: 36 adolescent/young adult participants
  Interventions: Other: Focus group

INTERVENTIONS:
Other: Working group — Participants will: 1) take a 10-min demographic survey; 2) join 3 x 60-min working group meetings in which they will review preliminary results, collaborate on curriculum design, and provide feedback; and 3) respond to prompts in 3 emails (approx 5-10 mins each).
  Groups: Working group members
Other: Focus group — Participants will take a 10-min demographic survey and join 1 x 30-min focus group meeting in which they will provide feedback on the curriculum in development.
  Groups: Focus group participants

SUMMARY:
The purpose of this study is to develop an electronic cigarette (e-cigarette) counter-marketing lesson for adolescents. The lesson will involve short videos designed to improve adolescents' cognition of e-cigarette marketing in the retail environment with the overall goal of reducing their susceptibility to use, intent to use, and actual use of e-cigarettes. Through this study, the study team will identify and refine the key messages that would make this lesson acceptable, feasible to implement, and effective in altering e-cigarette-related perceptions and potentially behaviors.

DETAILED DESCRIPTION:
This research comprises of 2 qualitative activities:

1. Working group: The study team will purposively invite a convenience sample of expert members (including middle/high school students, young adults, an educator, a parent, and curriculum design experts) to convene multiple times over several weeks (3 meetings via videoconference). The working group will convene to view preliminary results from formative research, collaborate on the development of this lesson curriculum, and otherwise offer meaningful input on study materials.
2. Focus groups: A convenience sample of adolescents/young adults will be enrolled to participate in a focus group via videoconferenc . Each participant will only participate in a single focus group. There will be ~4 participants in each focus group, and 9 focus groups overall. Before their focus group, each participant will complete a brief online survey that collects sociodemographics and outcome measures data. During their focus group, each participant will be asked to view and describe their opinion about broad counter-marketing strategies, messages, and participate in viewing mood-boards and video-storyboards using these messages. A trained facilitator will follow a standardized discussion guide to lead the focus groups.

These activities will occur sequentially over about 6 months. At the 6-month time point, the study team will have met the study's primary aim of having developed the e-cigarette counter-marketing lesson.

ELIGIBILITY:
WORKING GROUP MEMBERS

*Inclusion criteria

Youth participants:

* Middle school students may be 13-15 years
* High schoolers may be 16-18 years
* Young adults may be 19-29 years
* Provide a phone number for at least one backup contact (e.g, parent/guardian)

Curriculum design experts:

• Experience of at least 1 year in tobacco prevention or relevant public health field

Parent:

• Parent of a child who has e-cigarette use history or is currently using (preferred, but not essential)

Educator:

* Currently employed as teacher at a middle/high school All participants
* Provide their cell phone number and email address
* Fluent in English

  *Exclusion criteria
* Express inability to participate consistently across study working group meetings.

FOCUS GROUP PARTICIPANTS

*Inclusion criteria

* Adolescents and young adults ages 13-21 years
* Fluent in English
* Provide their cell phone number and email address
* Provide a phone number for at least one backup contact

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include individuals residing in the U.S. There will be 10 members of the expert working group (2 middle, 2 high school students, 2 young adults, 1 educator, 1 parent, and 4 curriculum design experts). There will be 36 adolescent and young adult participants of the focus groups.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Development of an e-cigarette counter-marketing lesson focused on the retail environment | At 6 months
  Key messages and message-delivery strategy will be developed, potentially comprising of short-form videos. The study team will ask working group members to rank draft messages and strategies for delivery in addition to eliciting qualitative information.

OTHER OUTCOMES:
Feasibility: Preferred recruitment advertisement | Baseline (pre-focus group)
  Self-reported data and/or qualitative data elicited from participants by prompting: Which Instagram advertisement made you interested to join this study?
Acceptability: Relevance to population(s) | During baseline focus group
  Qualitative data elicited from participants by prompting: How participants feel about relevance to and representation of age group and e-cigarette use status (e.g., "this message is not for me since I don't vape" or "I would not be interested," helpfulness of content to achieve different tobacco prevention goals such as raising awareness, prevention)
Acceptability: Desired improvements | During baseline focus group
  Qualitative data elicited from participants by prompting: How would you improve the messages? What changes would you make?
Perceived influence of content: Awareness | During baseline focus group
  Qualitative data elicited from participants by prompting: How helpful was it to include [key message in development] to raise awareness about e-cigarettes and e-cigarette marketing?
Perceived influence of content: Reducing appeal | During baseline focus group
  Qualitative data elicited from participants by prompting: How helpful was it to include [key message in development] to prevent adolescents from liking e-cigarette products?
Perceived influence of content: Purchase behaviors | During baseline focus group
  Qualitative data elicited from participants by prompting: How helpful was it to include [key message in development] to prevent/reduce e-cigarette purchase?
Perceived influence of content: Use prevention | During baseline focus group
  Qualitative data elicited from participants by prompting: How helpful was it to include [key message in development] to prevent/reduce adolescent e-cigarette use?
Feasibility: Device used to access lessons | During baseline focus group
  Qualitative data elicited from participants by prompting: Device most commonly used to access similar online/video content
Feasibility: Duration of engagement with components | During baseline focus group
  Average time in minutes to engage with draft messages, and study activities
E-cigarette use | Baseline (pre-focus group)
  A survey will ask participants, "Have you ever tried any of the following products, even one or two puffs?" (Yes/No). If "Yes," participants will see the question, "During the past 30 days, did you use any of the following products, even one or two puffs? (Yes/No)." If "Yes," participants will see the question, "On how many days out of the past 30 days, did you use a…" with a numeric response from 0-30 (drop-down option where participants could select only one response). If participants provided an answer from 1-30 to this question, the survey will ask, "In the past 7 days, on how many days did you use an e-cigarette or vape?" with a numeric response from 0-7 (drop-down option where participants could select only one response).
  (Products include:nicotine vape, THC (marijuana) vape, some kind of vape (don't know what was in it), cigarette, and nicotine pouch).
Susceptibility to Use E-cigarettes | Baseline (pre-Focus Groups)
  A survey will ask participants 4 questions adapted from the Enhanced susceptibility to smoking index, (1) "Have you ever been curious about e-cigarettes/vapes?; (2) "Do you think you will try an e-cigarette/vape in the next month?;" (3) Do you think you will try an e-cigarette/vape in the next year?; and (4) "If one of your best friends were to offer you an e-cigarette/vape, would you try it?" with responses on a 4-point Likert-type scale (Definitely yes; Probably yes; Probably not; and Definitely not). Across all 4 questions, any participant response except "Definitely not" will be classified as susceptible to using e-cigarettes.
Acceptability: Perceptions of anti-vaping educational content or counter-marketing | During focus groups
  The facilitator will ask participants about perceptions of anti-vaping ads, specifically inside and around retail stores
Marketing receptivity inside and around retail stores | At Baseline (pre-Focus groups) and During Baseline Focus Groups
  A survey and the focus group facilitator will ask about perceptions of e-cigarette brand recall among adolescents, appealing locations of advertising, ownership of merchandise, and receipt of free samples
Feedback on counter-marketing messages | During baseline focus groups
  The facilitator will ask participants: 1) Could you describe what was interesting or engaging? Probes: How would you improve what you just saw? What changes would you make? Comments on: a) individualized delivery; b) influencer-style; c) message? 2) Are there parts you would recommend excluding? Why? 3) How relevant was it to you? To people your age? 4) Was the language used easy to understand? 5) How does this messaging compare to what you have already seen? 6) How helpful was it to include the messages on marketing? a) raise awareness; b) prevent adolescents from liking products; c) prevent/ reduce e-cigarette purchase (in stores); d) prevent/ reduce e-cigarette purchase or sharing (with friends/family); and prevent/ reduce e-cigarette use? 7) If you were trying to prevent someone from starting to vape, what could be effective: a) aspects about vaping that you could bring up?; b) language that you could use?; c) images that you could use?; d) appeals that you could use?

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant survey data will be made available.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified data will be made available only after study publication (between 14-24 months after the end of the study).
Access Criteria: The Principal Investigator will provide data to those who indicate that they have received approval from an Institutional Review Board (IRB) or appropriate ethics committee, and execute a data use/sharing agreement.